CLINICAL TRIAL: NCT03370900
Title: Optimizing Skill Retention in Radiograph Interpretation: A Multicentre Randomized Control Trial
Brief Title: Learning Retention in Radiograph Interpretation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: New York University (Other); St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Kathy Boutis, Physician and Senior Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1000028986
Record Dates: First submitted 2017-12-02; First posted 2017-12-13 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2017-12

CONDITIONS: Fractures, Bone
Keywords: Education (Medical); Retention;
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: This was a four arm randomized control trial. All participants completed an 80-case deliberately practiced learning set of pediatric elbow radiographs followed by an immediate 20-case post-test. Following this, Group 1 had no testing until 12 months; Groups 2, 3, and 4 had testing (20 cases without feedback) every 2 months until 12 months, but Group 3 also had refresher education (20 cases with feedback) at six months while Group 4 had refresher education at two, six, and ten months.
Who Masked: Outcomes Assessor
Masking Description: All analyses were blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Learning and Assessment at 12 months (No Intervention): Study participants will complete an 80 case learning set followed by a 20-case post test. The study intervention in this group is a 20-case test at 12 months.
- Testing Every Two Months (Experimental): Study participants will complete an 80 case learning set followed by a 20-case post test. Study participants in this group will receive the following study interventions: 20-case post tests without any feedback at 2, 4, 6, 8, 10, 12 months.
  Interventions: Other: Testing
- Low Bolus Feedback (Experimental): Study participants will complete an 80 case learning set followed by a 20-case post test. Study participants in this group will receive the following study interventions: 20-case post tests at 2, 4, 6, 8, 10, 12 months. At 6 months, the 20-case post-test will be delivered with feedback.
  Interventions: Other: Testing
- High Bolus Feedback (Experimental): Study participants will complete an 80 case learning set followed by a 20-case post test. Study participants in this group will receive the following study interventions: 20-case post tests at 2, 4, 6, 8, 10, 12 months. At 4, 8, and 12 months, the 20-case post-test will be delivered with feedback.
  Interventions: Other: Testing

INTERVENTIONS:
Other: Testing — Participants either received 20 case testing with or without feedback
  Arms: High Bolus Feedback; Low Bolus Feedback; Testing Every Two Months

SUMMARY:
Learning retention after the deliberate practice of radiograph interpretation may be challenging for image types which are common enough to be clinically relevant but not so common that proficiency can be sustained through clinical practice. This is especially relevant for radiographs such as paediatric elbow films (EXR) that carry high risks for the patient if pathology is missed. Building on prior research in this area, this study will develop an innovative computer learning application for paediatric EXR interpretation. After an initial learning period, this study will quantitatively determine the rate of skill decay and the optimal timing for refresher-education.

DETAILED DESCRIPTION:
Objectives Learning retention after the deliberate practice of radiograph interpretation may be challenging for image types which are common enough to be clinically relevant but not so common that proficiency can be sustained through clinical practice. This is especially relevant for radiographs such as paediatric elbow films (EXR) that carry high risks for the patient if pathology is missed. Building on our prior research in this area, this study will develop an innovative computer learning application for paediatric EXR interpretation. After an initial learning period, this study will quantitatively determine the rate of skill decay and the optimal timing for refresher-education.

Design A prospective cohort design with purposive sampling will be used to develop the EXR education intervention. A four arm randomized control trial will be used to test for the outcomes of skill decay and optimal timing of refresher education.

Setting The education intervention will be developed at two tertiary care children's hospitals. Study participants will include physicians from two large paediatric education networks in the United States (Paediatric Outcomes in Simulation Education) and Canada (Paediatric Emergency Research Canada).

Statistical analysis For the primary analysis, a four-group multi-level model with time-points nested within participants will be used. Secondary analyses will include a time series approach within each block of 20 test EXR to check for sequential effects, and between each block to determine whether we can efficiently model skill decay curves that can separate the underlying learning attrition curve from the effects of "boluses" of education.

Conclusion This study anticipates that learners will increase their learning of elbow radiographs by participating in the deliberate practice of radiographs, with skill decay over time that will be mitigated by refresher education. The results will allow evidence based recommendations regarding refresher education for learning from item banks of radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and emergency medicine residents enrolled in an accredited residency in Canada and the United States

Exclusion Criteria:

* None

Max Age: 70 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 233 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Accuray | 12 months after learning intervention
  The percent of cases that were diagnosed correctly by the study participants

SECONDARY OUTCOMES:
Accuracy | 2, 4, 6, 8, 10 months
  The percent of cases that were diagnosed correctly by the study participants
Experience Curve | 12 months
  Learning and forgetting curve for each group by linking learning curve parameters (y-intercept, slope) with the amount of forgetting (T12 score).

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Boutis, Principal Investigator — The Hospital for Sick Children

IPD SHARING:
Plan to Share IPD: No